CLINICAL TRIAL: NCT07270627
Title: Cohorte Militaire et Son Exposome : étude Pilote rétrospective au Sein de la Population Des Sapeurs-pompiers (Actuellement en Exercice et Anciens Sapeurs-pompiers) de la Brigade Des Sapeurs Pompiers de Paris
Brief Title: French Military Firefighters to Assess Relationships Between Exposome and Health.
Acronym: COMITEX-BSPP
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023PBMD02
Record Dates: First submitted 2025-09-10; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Health Adult Subjects; Exposure Occupational; Health Behavior, Risky; Occupational Health; Exposure; Firefighters; Military Personnel; Observational Study
Keywords: Occupational exposure; health; military; exposome; occupational
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active-duty firefighters (military): Active-duty firefighters who will be considered several subgroups according exposure studied.
- Veteran firesoldiers: Veteran firesoldiers who will partitioned in several subgroups according exposure studied.

SUMMARY:
The aim of the study is to describe professional exposures and health events among French military firefighters (both active-duty personnel and veterans) and identify potential relationships between the exposome (the total history of occupational and personal exposures) and health status in these populations. The study is based on a self-administered questionnaire that collects retrospective and present information about exposures and health conditions.

DETAILED DESCRIPTION:
This group of military personnel is professionally exposed, in the diversity of its activities (rescue of victims but also firefighting, protection of property, technological risks, traffic accidents, assistance to individuals, etc.), to multiple health risks, as specified in a report by ANSES (ANSES 2019):

* chemical and particulate substances (polycyclic aromatic hydrocarbons (PAHs) present in fire smoke in particular, asbestos, diesel emissions);
* biological agents (viruses, bacteria, mold, etc.) or physical agents (noise, ionizing or non-ionizing radiation such as electromagnetic fields, optical radiation, radioactivity, extreme temperatures and pressures, vibrations, etc.);
* organizational constraints (time constraints, intensity and pace of work) and psychosocial constraints, including exposure to violence.

Furthermore, in 2007, the International Agency for Research on Cancer (IARC) classified firefighting as "probably carcinogenic to humans" based on limited evidence of cancer in humans, particularly non-Hodgkin's lymphoma, prostate cancer, and testicular cancer (IARC 2007). In 2022, occupational exposure of firefighters was considered "carcinogenic to humans" based on sufficient evidence for mesothelioma and bladder cancer and limited evidence for colon, prostate, and testicular cancers, melanoma, and non-Hodgkin's lymphoma (IARC 2022, Senate 2024).

A study conducted within the BSPP would not only provide better documentation of the impact of the military firefighting profession on health, but also estimate the feasibility of such a study: participation and adherence rates to the cohort, acceptability of the inclusion questionnaire and the questions asked with feedback. The data collected in the questionnaires that accompany nationwide cohort studies are indeed substantial, with a wide variety of questions requiring memory recall. Consequently, the choice and structure of the questions asked are essential in order to minimize the amount of missing data (non-response bias) and maintain a satisfactory quality of data collection, thereby ensuring the internal and external validity of the results obtained. The study among active and former firefighters will thus validate the method chosen to include participants in the future general military cohort, as well as the initial questionnaire. At the end of the questionnaire, questions about the participants' experience will be asked in order to assess the acceptance and feasibility of a future study.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty or veteran military personnel from French Paris firefighter brigade.
* Aged at least 18.
* Not opposed to participate to the study

Exclusion Criteria:

* Opposition to participate
* veterans under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active-duty personnel from Paris firefighters brigade as a whole. Veterans from Paris firefighters brigade with known email address.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To identify associations between occupational and environnment exposures and the health status reported by current and former military firefighters, | Period at enrollment in the study (from January 2026 to March 2026) of Health outcome (with retrospective assessment of exposure in the past as firefighter).
  To identify associations between occupational and environnment exposures and the health status reported by current and former military firefighters, through difference in prevalence of the health events (muscoskelatal, psychologic, cardiovascular... ) studied between those exposed to one or more risk factors (chemical/ physical/ psychological) and those not exposed to these factors.

IPD SHARING:
Plan to Share IPD: No
(security and regulation)